CLINICAL TRIAL: NCT03969121
Title: A Phase III Randomized, Double-Blind, Neoadjuvant Study of Hormonal Therapy Plus Palbociclib Versus Hormonal Therapy Plus Placebo in Women With Operable, Hormone Sensitive and HER2-Negative Primary Breast Cancer
Brief Title: Neoadjuvant Hormonal Therapy Plus Palbociclib in Operable, Hormone Sensitive and HER2-Negative Primary Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyoto Breast Cancer Research Network (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OOTR-N016/KBCRN-B-003/HT-PAB
Record Dates: First submitted 2019-05-13; First posted 2019-05-31 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2021-06

CONDITIONS: Breast Cancer Female; Hormone Receptor Positive Malignant Neoplasm of Breast
Keywords: Palbociclib; Breast Cancer; PEPI
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo + Endocrine therapy (Active Comparator): Endocrine therapy for 16 weeks plus placebo
  Interventions: Drug: Endocrine therapy
- Palbociclib + Endocrine therapy (Active Comparator): Endocrine therapy for 16 weeks plus Palbociclib
  Interventions: Drug: Palbociclib; Drug: Endocrine therapy

INTERVENTIONS:
Drug: Palbociclib — Palbociclib will be administered orally once a day for 21 days every 28-day cycle followed by 7 days off treatment
  Arms: Palbociclib + Endocrine therapy
Drug: Endocrine therapy — Pre- and peri-menopausal women will be receiving Ovarian Function Suppression (OFS) by either leuprorelin subcutaneous 3.75 mg q28days or goserelin subcutaneous 3.6 mg q28days plus tamoxifen 20 mg QD in 28-day cycles. Post-menopausal women will receive letrozole 2.5 mg QD in 28-day cycles.

SUMMARY:
The study is a randomized, double blind, placebo controlled, Phase 3 clinical trial with the primary objective of demonstrating the efficacy of palbociclib in combination with Endocrine therapy over Endocrine therapy alone measured by PEPI and EndoPredict™ EPclin Score in women with operable HR+, HER2 negative breast cancer . The Clinical Response Rate, drop in Ki67 index ≤ 2.7% and Breast conserving rate will be compared between two arms.

ELIGIBILITY:
Inclusion Criteria:

1. Pre/peri- or post-menopausal women 18 years and older (or local legal age, whichever is higher)
2. Primary tumor greater than 15 mm in diameter
3. Histologically proven invasive breast cancer
4. Positive hormone receptor (ER and/or PgR ≥1% in proportion of positive staining score)
5. Negative HER-2 receptor (based on 2018 ASCO/CAP Guideline)
6. Ki67 index equal to or greater than 14% (Ki67 ≥ 14%) by central assessment using actual or virtual slides
7. Eastern Cooperative Oncology Group Performance Status (ECOG PS) ≤ 1
8. No previous history of radiotherapy or systemic therapy including chemotherapy and hormone therapy for breast cancer
9. Laboratory values must be as follows:

   Absolute neutrophil count: ≥ 1,500/mm3

   Platelets: ≥ 100,000/mm3

   Hemoglobin: ≥ 9 g/dL

   Bilirubin: ≤ 1.5 × upper limits of normal (ULN)

   Serum Creatinine: ≤ 1.5 × ULN

   Alkaline phosphatase: ≤ 2 × ULN

   AST and ALT: ≤ 2 × ULN

   Cardiac function: Normal finding of Electrocardiogram (ECG) QTc ≤ 480 msec (based on the mean value of the triplicate ECGs).
10. Able to give written informed consent form
11. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria:

1. Male
2. Locally advanced breast cancer ( Any T4 or Any N2, N3), or distant metastasis
3. Multicentric breast cancer (Note: Multifocal breast cancer,located in one quadrant/are is eligible)
4. Prior treatment with chemotherapy, radiotherapy and/or endocrine therapy
5. Previous use of SERMs such as raloxifene.
6. Prior therapy with any CDK4/6 inhibitor or with everolimus, or any agent whose mechanism of action is to inhibit the PI3K-mTOR pathway.
7. Prior history of other malignancy within 5 years of study entry, aside from basal cell carcinoma of the skin or carcinoma-in-situ of the uterine cervix
8. Major surgery within 3 weeks of first study treatment
9. Patients treated within the last 7 days prior to randomization with:

   * Food or drugs that are known strong and moderate CYP3A4 inhibitors (e.g., amprenavir, aprepitant, atazanavir, boceprevir, casopitant, cimetidine, ciprof-loxacin, clarithromycin, conivaptan, cobicistat, crizotinib, cyclosporine, da-runavir, diltiazem, dronedarone, elvitegravir, erythromycin, fluconazole, fosamprenavir, imatinib, indinavir, isavuconazole, istradefylline, itraconazole,ketoconazole, letermovir, lopinavir, mibefradil, miconazole, nefazodone, nelfinavir, nilotinib, posaconazole, ritonavir, saquinavir, schisandra sphenan-thera extract, telaprevir, telithromycin, tofisopam, verapamil, voriconazole, and grapefruit, grapefruit juice or any product containing grapefruit);
   * Drugs that are known strong and moderate CYP3A4 inducers (e.g., bosentan, carbamazepine, efavirenz, etravirine, modafinil, phenobarbital, phenytoin, ri-fampin, rifapentin, and St. John's wort);
10. Any of the following in the previous 6 months of randomization: myocardial in-farction, severe/unstable angina, ongoing cardiac dysrhythmias of NCI CTCAE version 4.03 grade ≥ 2, atrial fibrillation of any grade, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident in-cluding transient ischemic attack, or symptomatic pulmonary embolism
11. Family or personal history of long or short QT syndrome, Brugada syndrome or known history of QTc prolongation, or Torsade de Pointes (TdP).
12. Uncontrolled electrolyte disorders (eg, hypocalcemia, hypokalemia, hypomag-nesemia) that can compound the effects of a QTc-prolonging drug.
13. Active inflammatory bowel disease or chronic diarrhea. Short bowel syndrome. Upper gastrointestinal surgery including gastric resection.
14. Prior hematopoietic stem cell or bone marrow transplantation.
15. Known abnormalities in coagulation such as bleeding diathesis, or treatment with anticoagulants precluding subcutaneous injections of leuprorelin or goserelin.
16. Hepatitis B and/or hepatitis C carriers (Patients with HBsAg+ or HBV-DNA+ who need antiviral treatment during any anti-cancer therapy based on guidelines are excluded even if the patient's hepatic function is normal. Patients with HCVAb+, whose HCV-RNA is positive (+) are excluded.)
17. Known human immunodeficiency virus (HIV) infection
18. Known hypersensitivity to anti-aromatase drugs, tamoxifen or any cell cycle in-hibitor.
19. Patients who are pregnant or lactating. Patients of childbearing potential and/or her partner who are unwilling or unable to use a method of highly effective non-hormonal contraception throughout the study and continue for at least 21 days in patients after the last dose of investigational drug.
20. Other severe acute or chronic medical or psychiatric condition, or laboratory ab-normality that would impart, in the judgment of the investigator, excess risk as-sociated with study participation or study drug administration, or which, in the judgment of the investigator, would make the patient inappropriate for entry into this study
21. Patients who are investigational site staff members or relatives of those site staff OOTR-N016/KBCRN-B-003/HT-PAB Protocol (version 1.2 dated Oct 11, 2018) 24 members or patients who are the sponsor employees directly involved in the con-duct of the trial.
22. Participation in other studies involving investigational drug (s) (Phases 1-4) within 2 weeks before randomization and/or until a visit at 4 weeks (+7 days) after operation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
Pre-operative Endocrine Prognostic Index (PEPI Score) | 4 months
  The PEPI score is derived from four factors assigned a numerical score following neoadjuvant endocrine therapy, ( including Ki67 expression in the surgical specimen, pathologic tumor size, lymph node status, and estrogen receptor (ER) level).
  The PEPI score is the sum of each component score and shows the risk points for relapse-free survival. PEPI=0 means low risk. PEPI= 1 to 3 means intermediate risk .
  PEPI more than 4 means high risk.
EndoPredict™ EPclin Score | 4 months
  EndoPredict is a multigene test used to predict the risk of distant recurrence of early stage, ER positive ,HER-2 Negative invasive breast cancer. EndoPredict Clinical Score (EP clin ) categorizes patinets into low and high risk groups.Combination of the 12-Gene Molecular Score, tumor stage and lymph node status, generating an EPclin Risk Score.The EPclin Risk Score is calculated, according to the model, as:
  EPclin Risk Score = (0.35 * tumor size) + (0.64 * lymph node status) + (0.28 * 12-Gene Molecular Score) EPclin Risk Scores from 1.0 through 3.3 shows low risk of recurrencein 10 years.EPclin Risk Scores from 3.4 through 6.0 shows high risk of recurrence in 10 years.

SECONDARY OUTCOMES:
Clinical Response Rate | 4 months
  Observing any reduction in largest tumor diameter on clinical breast examination and ultrasound imaging of breast and axilla after 4 months
Ki67 change | 4 months
  Drop in Ki67 index to less than or equal to 2.7%
pathological response rate | 4 months
  Evaluating the rate of pathological Complete Response based on assessment of surgical specimen
Breast conserving rate | 4 months
  Calculating the rate of breast conserving surgery based on the number of each surgery type
Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment as Assessed by CTCAE v4.03 | 4 months
  Type, incidence, severity (as graded by National Cancer Institute - Common Terminology Criteria for Adverse Events [NCI CTCAE] v4.03), seriousness and relationship to study medications of adverse events (AE) and any laboratory abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: Masakazu Toi, MD,PhD, Principal Investigator — Kyoto University, Professor of Breast Surgery Department; Louis WC Chow, MD,PhD, Principal Investigator — Organisation for Oncology and Translational Research (OOTR); Takayuki Ueno, MD,PhD, Principal Investigator — Cancer Institute Hospital of JFCR, Department Director, Breast Surgical Oncology Department
Locations (25):
- Australia (2):
  - Monash Health, Clayton
  - Peter MacCallum Cancer Centre, Melbourne
- UNIMED Medical Institute, Hong Kong, Hong Kong
- Japan (14):
  - Amagasaki General Medical Center, Amagasaki, Hyōgo
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Kyushu Cancer Center, Fukuoka
  - Sagara Hospital, Kagoshima
  - Kobe City Medical Center General Hospital, Kobe
  - Kyoto University Hospital, Kyoto
  - Aichi Cancer Center, Nagoya
  - Tazuke Kofukai, Medical Research Institute, Kitano Hospital, Osaka
  - Saitama Cancer Center, Saitama
  - Toranomon Hospital, Tokyo
  - Tokyo Metropolitan Komagome Hospital, Tokyo
  - Cancer Institute Hospital Of JFCR, Tokyo
  - Kyorin University Hospital, Tokyo
  - Kanagawa Cancer Center, Yokohama
- South Korea (4):
  - National Cancer Center, Korea, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam
  - Korea Cancer Center Hospital, Seoul
  - Seoul National University College of Medicine, Seoul
- Taiwan (4):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
  - Sun Yat-Sen Cancer Center, Taipei

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ueno T, Chow LWC, Han W, Huang CS, Mann GB, Morita S, Haga H, Fakhrejahani E, Kobayashi T, Bando H, Inoue K, Tokiwa M, Suwa H, Aruga T, Minamiguchi S, Yamada Y, Tanabe Y, Takada M, Yamashita T, Iwata H, Chung CF, Takahara S, Tokunaga E, Imoto S, Lee ES, Sagara Y, Kim JH, DeBoer RH, Kim HA, Lai HW, Hou MF, White M, Umeyama Y, Toi M. Neoadjuvant palbociclib in women with operable, hormone receptor-positive breast cancer. Endocr Relat Cancer. 2025 Sep 11;32(9):e240353. doi: 10.1530/ERC-24-0353. Print 2025 Sep 1. PMID 40888443